CLINICAL TRIAL: NCT01242748
Title: An Open-label, Multi-Centre, Extension Trial, Evaluating the Long-Term Progression-Free Survival of Degarelix or Goserelin Three-Month Dosing Regimens in Patients With Prostate Cancer Requiring Androgen Deprivation Therapy
Brief Title: A Degarelix Trial in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate recruitment resulting in a too low patient number for collection of long term efficacy data.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS35A; 2010-021434-55 (EudraCT Number)
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Degarelix 240 mg/480 mg (Experimental)
  Interventions: Drug: Degarelix
- Goserelin acetate (Active Comparator)
  Interventions: Drug: Goserelin acetate

INTERVENTIONS:
Drug: Degarelix — The degarelix doses were administered by subcutaneous (s.c.) injections into the abdominal wall. In the main CS35 trial, a starting dose of 240 mg degarelix was administered on Day 0. One month later a maintenance dose of 480 mg was administered. This was repeated after 4, 7, and 10 months (ie a total of 5 administrations in the main trial). In the CS35A extension trial, the participants received the same treatment as in the main trial ie the degarelix treated participants continued to receive degarelix 480 mg s.c. treatment every three months.
  Other Names: Firmagon; FE200486
  Arms: Degarelix 240 mg/480 mg
Drug: Goserelin acetate — The goserelin doses were administered by subcutaneous (s.c.) implants into the abdominal wall. In the main CS35 trial, an initial dose of 3.6 mg goserelin was administered on Day 0. One month later a subsequent dose of 10.8 mg was administered and this was repeated after 4, 7, and 10 months (ie a total of 5 implants in the main trial). In the CS35A extension trial, the participants received the same treatment as in the main trial ie the goserelin treated participants continued to receive goserelin acetate 10.8 mg s.c. implants every three months.
  Other Names: Zoladex
  Arms: Goserelin acetate

SUMMARY:
A phase III extension trial comparing the efficacy and safety of degarelix 3 month depot with the established therapy Zoladex 3 month implant in patients with prostate cancer.

DETAILED DESCRIPTION:
CS35A was an open-label, multicentre, comparative non-inferiority extension trial to the Phase 3 CS35 trial (NCT00946920).

In the main CS35 trial, participants were randomised 2:1 to treatment with degarelix or goserelin, respectively. All participants who completed the main CS35 trial after initiation of the CS35A trial were eligible to enrol into this extension trial, provided that their treatment could continue uninterrupted. Patients entering the CS35A trial continued with the same 3-monthly treatment as they received in CS35 (i.e. degarelix 480 mg or goserelin 10.8 mg).

It was intended that patients enrolled in the CS35A trial would receive treatment with degarelix or goserelin at 3-month intervals for a period of 40 months (including 13 months' treatment in CS35). It was, however, decided to prematurely terminate the CS35A trial due to an insufficient number of patients being enrolled. Maximum exposure of treatment was 111 weeks (in both treatment arms).

The baseline characteristics are based on the CS35A Full Analysis Set (FAS)defined as all participants who received at least one dose of degarelix or goserelin acetate during CS35A and had at least one efficacy assessment after dosing. All efficacy analyses were performed for the CS35/CS35A FAS defined as all participants who received at least one dose of degarelix or goserelin acetate during CS35 and had at least one efficacy assessment after dosing. All safety analyses were performed for the CS35/CS35A Safety analysis set, which included all patients who received at least one dose of degarelix or goserelin acetate during CS35.

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent prior to any trial-related activity is performed. (A trial-related activity is defined as any procedure that would not have been performed during the normal management of the patient).
* Has completed the CS35 trial.

Exclusion Criteria:

* Has been withdrawn from the CS35 trial.
* Has had end of trial visit in CS35 prior to approval of the CS35A protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (63):
- United States (8):
  - University of Colorado School of Medicine, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Urology Associates of Dover, PA, Dover, Delaware
  - South Florida Medical Research, Aventura, Florida
  - Urology Group of New Mexico, PC, Albuquerque, New Mexico
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio Research, Pa, San Antonio, Texas
  - Seattle Urology Research Center, Burien, Washington
- AZ Groeninge - Campus Sint-Maarten, Kortrijk, Belgium
- Canada (5):
  - Jonathan Giddens Medicine Professional Corporation, Brampton, Ontario
  - Southern Interior Medical Research Inc., Kelowna
  - Mor Urology, Inc., Newmarket
  - Investigational site, Scarborough
  - Investigational site, Toronto
- Czechia (6):
  - Urocentrum Brno, Brno
  - Nemocnice Jindrichuv Hradec, a.s., Jindřichův Hradec
  - Kromerizska nemocnice a.s., Kroměříž
  - Fakultni nemocnice v Motole, Praha 5, Prague
  - Vseobecna fakultni nemocnice v Praze, Praha 2, Prague
  - Krajska nemocnice T. Bati a.s., Zlín
- Finland (3):
  - ODL Terveys Oy, Oulu
  - Pohjois-Karjalan keskussairaala, Tampere
  - Tampereen yliopistollinen sairaala, Tampere
- Germany (2):
  - Gemeinschaftspraxis Rudolph & Wörner, Kirchheim
  - Urologische Studienpraxis, Nürtingen
- Hungary (9):
  - Fövárosi Önkormányzat Bajcsy-Zsilinszky Kórház, Budapest
  - Fövárosi Önkormányzat uzsoki utcai Kórház, Budapest
  - Semmelweis Egyetem, Budapest
  - Dombóvári Szent Lukács Egészségügyi Nonprofit Kft., Dombóvár
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Miskolci Semmelweis Ignác Egészségügyi Központ és Egyetemi Oktató Kórház Nonprofit Kft, Miskolc
  - Pécsi Tudományegyetem, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Jávorszky Ödön Kórház, Vác
- Mexico (6):
  - Hospital Christus Muguerza del Parque, Chihuahua, Chih.
  - Hospital Angeles Culiacan, Culiacan, Sinaloa
  - Consultorio de Especialidad en Urologia Privado, Durango
  - Médica Sur, S.A.B. de C.V., Mexico City
  - Hospital Angeles Lindavista, Mexico City, DF
  - Consultorio Medico, Zapopan, Jalisco
- Netherlands (2):
  - Catharina-ziekenhuis, Eindhoven
  - MC Haaglanden, The Hague
- Poland (3):
  - SPZOZ Wojewodzki Szpital Zespolony im. J.Sniadeckiego, Bialystok
  - Centrum Medyczne Medur Sp. z o.o., Bielsko-Biala
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku, Słupsk
- Romania (10):
  - Private Medical Center SRL, Arad
  - Brasov Emergency Clinical County Hospital, Brasov
  - "Prof. Dr. Th. Burghele" Clinical Hospital, Bucharest
  - "Sfantul Ioan" Emergency Clinical Hospital, Bucharest
  - Dinu Uromedica, Bucharest
  - Fundeni Clinical Institute of Uronephrology and Renal Transplantation, Bucharest
  - PROVITA 2000 Medical Center, Constanța
  - "Dr. C.I. Parhon" Clinical Hospital, Iași
  - Vita Care Flav Medical Center, Piteşti
  - Sibiu Emergency Clinical County Hospital, Sibiu
- Ukraine (6):
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Donetsk Regional Clinical Territorial Medical Association, Donetsk
  - Regional Clinical Center of Urology and Nephrology n.a. V.I.Shapoval, Kharkiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Odesa Regional Clinical Hospital, Odesa
  - Municipal Institution "Zaporizhzhia Regional Clinical Hospital", Zaporizhzhya
- United Kingdom (2):
  - Ipswich Hospital, Ipswich
  - The Royal Marsden NHS Foundation Trust, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who completed the main CS35 trial after initiation of the CS35A extension trial were eligible to enrol into CS35A.
Pre-assignment Details: Participants entering the CS35A trial continued with the same 3-monthly treatment as they received in CS35 (i.e. degarelix 480 mg or goserelin 10.8 mg).
Period: Overall Study
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Started | 194 (Enrolled in CS35A, CS35A Full Analysis Set.) | 94
CS35/CS35A Safety Analysis Set | 565 (Received at least 1 dose of trial drug during the main CS35 trial.) | 283
CS35/CS35A Full Analysis Set (FAS) | 565 (Received at least 1 dose of trial drug during CS35+had at least 1 efficacy assessment after dosing.) | 282
Completed | 156 (These participants were ongoing when the trial was closed by the Sponsor.) | 80
Not Completed | 38 | 14
Not completed — Adverse Event | 10 | 5
Not completed — Lost to Follow-up | 6 | 2
Not completed — Physician Decision | 3 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Miscellaneous reasons | 8 | 3

BASELINE CHARACTERISTICS:
Population: CS35A Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate | Total
Number analyzed (Participants) | 194 | 94 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (8.4) | 71.3 (7.0) | 72.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 194 | 94 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 34 | 21 | 55
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 154 | 68 | 222
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Median Baseline Serum Testosterone Levels [Median (Full Range); unit: nanogram per milliliter (ng/mL)] | 4.41 [0.68 to 13.3] | 4.65 [1.55 to 13.2] | 4.52 [0.68 to 13.3]
Median Baseline Serum Prostate-specific Antigen Levels [Median (Full Range); unit: ng/mL] | 20.6 [0.4 to 8762] | 16.6 [1.49 to 12961] | 18.7 [0.4 to 12961]

OUTCOME MEASURES:

1. Primary Outcome: Hazard Ratio of Prostate-specific Antigen (PSA) Progression-free Survival (PFS) Failure Rates During 3 Years' Treatment Between Degarelix and Goserelin
Description: PSA PFS failure is defined as either PSA failure (defined as increase in serum PSA of 50%, and at least 5 ng/mL, compared to nadir, measured on two consecutive occasions at least 2 weeks apart) or death, whichever is first. The number below present the unadjusted rates (estimated using the Kaplan-Meier method) of no PSA-PFS.
Time Frame: From baseline to 3 years
Population: CS35 (NCT00946920)/CS35A Full Analysis Set (degarelix n=565; goserelin n=282). The analysis population was pre-specified in the study protocol and statistical analysis plan.
Measure: Number (95% Confidence Interval); unit: percentage of no PSA-PFS
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percentage of no PSA-PFS | 75.5 [69.1 to 80.7] | 75.4 [64.5 to 83.4]
Statistical Analysis 1: Comparison: Degarelix 240 mg/480 mg vs Goserelin Acetate; The hazard ratio of PSA PFS failure rates was estimated using the Cox proportional hazard model with time to PSA PFS failure as dependent and treatment as independent variables and adjusted for baseline PSA category, prostate cancer stage, weight and geographical region. Degarelix was to be considered non-inferior to goserelin if the upper limit of the two-sided 95% confidence interval (CI) of the adjusted hazard ratio was less than or equal to the non-inferiority margin of 1.33; Test type: Non-Inferiority or Equivalence — Degarelix was considered to be non-inferior to goserelin with regard to the hazard ratio of PSA PFS failure rates as the upper limit of the two-sided 95% CI of the adjusted hazard ratio was less than the non-inferiority margin of 1.33; p = 0.1589, Cox proportional hazard model; Hazard Ratio (HR) = 0.774, 95% CI 2-sided [0.542 to 1.106]

2. Secondary Outcome: Hazard Ratio of PFS Failure Rates During 3 Years Treatment Between Degarelix and Goserelin
Description: PFS failure is defined as either PSA failure, introduction of additional therapy related to prostate cancer (radiation, anti-androgens or second-line treatment), or death, whichever is first. The number below present the unadjusted rates (estimated using the Kaplan-Meier method) of no PFS failure.
Time Frame: From baseline to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of no PFS failure
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percentage of no PFS failure | 71.5 [66.0 to 76.2] | 69.0 [58.0 to 77.7]
Statistical Analysis 1: Comparison: Degarelix 240 mg/480 mg vs Goserelin Acetate; The hazard ratio was estimated using the Cox proportional hazard model; Test type: Superiority or Other; p = 0.1244, Cox proportional hazard model; Hazard Ratio (HR) = 0.783, 95% CI 2-sided [0.574 to 1.070]

3. Secondary Outcome: Hazard Ratio of PSA Failure Rates During 3 Years Treatment Between Degarelix and Goserelin
Description: PSA failure is defined as increase in serum PSA of 50%, and at least 5 ng/mL, compared to nadir, measured on two consecutive occasions at least 2 weeks apart. The number below present the unadjusted rates (estimated using the Kaplan-Meier method) of no PSA failure.
Time Frame: From baseline to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of no PSA failure
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percentage of no PSA failure | 77.5 [71.0 to 82.7] | 79.6 [68.9 to 86.9]
Statistical Analysis 1: Comparison: Degarelix 240 mg/480 mg vs Goserelin Acetate; The hazard ratio was estimated using the Cox proportional hazard model; Test type: Superiority or Other; Hazard Ratio (HR) = 0.856, 95% CI 2-sided [0.580 to 1.263]

4. Secondary Outcome: Hazard Ratio of Testosterone Escape Rates During 3 Years' Treatment Between Degarelix and Goserelin
Description: Testosterone escape is defined as serum levels >0.5 ng/mL. The number below present the unadjusted rates (estimated using the Kaplan-Meier method) of no testosterone escape.
Time Frame: From baseline to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of no testosterone escape
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percentage of no testosterone escape | 83.7 [77.4 to 88.4] | 96.7 [93.7 to 98.2]
Statistical Analysis 1: Comparison: Degarelix 240 mg/480 mg vs Goserelin Acetate; The hazard ratio was estimated using the Cox proportional hazard model; Test type: Superiority or Other; p = 0.0005, Cox proportional hazard model; Hazard Ratio (HR) = 3.511, 95% CI 2-sided [1.739 to 7.090]

5. Secondary Outcome: Hazard Ratio of the Rates of Introduction of Additional Therapy Related to Prostate Cancer During 3 Years' Treatment Between Degarelix and Goserelin
Description: Additional therapy related to prostate cancer included radiation, anti-androgens and second-line treatment. The number below present the unadjusted rates (estimated using the Kaplan-Meier method) of no additional therapy related to prostate cancer.
Time Frame: From baseline to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of no additional therapy
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percentage of no additional therapy | 84.5 [80.0 to 88.1] | 83.4 [77.3 to 88.0]
Statistical Analysis 1: Comparison: Degarelix 240 mg/480 mg vs Goserelin Acetate; The hazard ratio was estimated using the Cox proportional hazard model; Test type: Superiority or Other; p = 0.143, Cox proportional hazard model; Hazard Ratio (HR) = 0.739, 95% CI 2-sided [0.493 to 1.108]

6. Secondary Outcome: Hazard Ratio of Mortality Rates During 3 Years' Treatment Between Degarelix and Goserelin
Description: The number below present the unadjusted rates (estimated using the Kaplan-Meier method) of death.
Time Frame: From baseline to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of deaths
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percentage of deaths | 4.6 [2.4 to 8.5] | 5.3 [2.6 to 10.5]
Statistical Analysis 1: Comparison: Degarelix 240 mg/480 mg vs Goserelin Acetate; The hazard ratio was estimated using the Cox proportional hazard model; Test type: Superiority or Other; p = 0.2212, Cox proportional hazard model; Hazard Ratio (HR) = 0.595, 95% CI 2-sided [0.259 to 1.368]

7. Secondary Outcome: Serum Levels of Testosterone During 3 Years' Treatment With Degarelix or Goserelin
Description: Median testosterone levels are presented as absolute values in nanograms per milliliter (ng/mL) at baseline and after 1, 6, 12, 19, and 22 months. One month equals 28 days. After 22 months, only a limited number of samples were analysed.
Time Frame: Baseline and after 1, 6, 12, 19, and 22 months
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
ng/mL
  Baseline | 4.52 [0.56 to 14.5] | 4.62 [0.07 to 13.2]
  Month 1 | 0.10 [0.015 to 3.85] | 0.16 [0.04 to 1.77]
  Month 6 | 0.09 [0.015 to 1.57] | 0.09 [0.015 to 0.32]
  Month 12 | 0.10 [0.015 to 1.1] | 0.09 [0.015 to 0.44]
  Month 19 | 0.11 [0.05 to 2.22] | 0.05 [0.05 to 0.43]
  Month 22 | 0.11 [0.05 to 3.4] | 0.05 [0.05 to 0.23]

8. Secondary Outcome: Serum Levels of Prostate-specific Antigen (PSA) During 3 Years' Treatment With Degarelix or Goserelin
Description: Median PSA levels are presented as absolute values in nanograms per milliliter (ng/mL) at baseline and after 1, 6, 12, 19, and 22 months. One month equals 28 days. After 22 months, only a limited number of samples were analysed.
Time Frame: Baseline and after 1, 6, 12, 19, and 22 months
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
ng/mL
  Baseline | 19 [0.26 to 8762] | 19.1 [0.005 to 12961]
  Month 1 | 3.79 [0.03 to 1540] | 6.5 [0.005 to 645]
  Month 6 | 0.82 [0.005 to 2648] | 0.73 [0.005 to 607]
  Month 12 | 0.6 [0.005 to 6889] | 0.43 [0.005 to 1802]
  Month 19 | 0.54 [0.005 to 712] | 0.28 [0.005 to 1150]
  Month 22 | 0.535 [0.005 to 252] | 0.26 [0.005 to 646]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signed informed consent until the last visit (maximum 111 weeks of treatment).
Description: Adverse events were evaluated at each visit. The analysis population was the CS35/CS35A (NCT00946920)/CS35A Safety Analysis Set (degarelix n=565; goserelin n=283). The analysis population was pre-specified in the study protocol and statistical analysis plan.
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Serious Adverse Events (participants affected / at risk) | 58/565 | 33/283
Other Adverse Events (participants affected / at risk) | 430/565 | 197/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 240 mg/480 mg (N=565) | Goserelin Acetate (N=283)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Blindness transient (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Sudden death (General disorders) | 3 | 0
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour local invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 240 mg/480 mg (N=565) | Goserelin Acetate (N=283)
Injection site pain (General disorders) | 174 | 4
Injection site erythema (General disorders) | 123 | 0
Injection site nodule (General disorders) | 52 | 0
Fatigue (General disorders) | 27 | 15
Pyrexia (General disorders) | 31 | 8
Injection site swelling (General disorders) | 36 | 0
Oedema peripheral (General disorders) | 13 | 16
Urinary tract infection (Infections and infestations) | 26 | 18
Weight increased (Investigations) | 27 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 23
Hot flush (Vascular disorders) | 161 | 76
Hypertension (Vascular disorders) | 23 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.